CLINICAL TRIAL: NCT04051463
Title: Prospective Randomized Study to Determine Whether Use of Rhopressa™ Can Ameliorate Corneal Edema Associated With Fuchs Dystrophy
Brief Title: Rhopressa for Corneal Edema Associated With Fuchs Dystrophy
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Price Vision Group (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2019-007
Record Dates: First submitted 2019-08-07; First posted 2019-08-09 (Actual); Results first posted 2021-09-24 (Actual); Last update posted 2021-10-19 (Actual); Status verified 2021-09

CONDITIONS: Fuchs Endothelial Dystrophy
MeSH Terms: conditions — Fuchs' Endothelial Dystrophy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The active drug and placebo will be provided in 2.5 ml bottles identical, in appearance. Only the designated dosing coordinator is unmasked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Netarsudil (Active Comparator): A drop of Netarsudil 0.02% ophthalmic solution will be instilled into both eyes once daily at night.
  Interventions: Drug: Netarsudil Ophthalmic Solution
- Placebo (Placebo Comparator): A placebo eye drop, consisting of the vehicle for netarsudil ophthalmic solution without the active ingredient, will be instilled into both eyes once daily at night.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Netarsudil Ophthalmic Solution — Netarsudil eye drops instilled once daily
  Other Names: Rhopressa
  Arms: Netarsudil
Drug: Placebo — Placebo eye drops instilled once daily
  Other Names: Rhopressa vehicle without active ingredient
  Arms: Placebo

SUMMARY:
The study objective is to determine whether use of Rhopressa improves the ability of corneal endothelial cells to maintain appropriate corneal hydration in patients with Fuchs endothelial corneal dystrophy (FECD), which could help delay or prevent the need for a corneal transplant.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Male or female patient diagnosed with FECD and corneal edema evident by slit lamp exam and/or corneal tomography.
* Patient is able and willing to administer eye drops.
* Patient is able to comprehend and has signed the Informed Consent form.

Exclusion Criteria:

* Active intraocular inflammation, corneal ulceration, keratitis, or conjunctivitis.
* Known sensitivity to any of the ingredients in the study medications.
* Abnormal eyelid function.
* History of herpetic keratitis.
* History of non-compliance with using prescribed medication.
* Current or planned pregnancy within the study duration.
* Concurrent involvement or participation in another randomized clinical trial within 30 days prior to enrollment in this study.
* Any ocular or systemic condition (i.e., UNCONTROLLED systemic disease) or situation which in the investigator's opinion may put the patient at significant risk, confound the study results, or interfere significantly with the patient's participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2019-08-05 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francis W Price, Jr, MD, Principal Investigator — Price Vision Group
Locations (1):
- Price Vision Group, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Price MO, Price FW Jr. Randomized, Double-Masked, Pilot Study of Netarsudil 0.02% Ophthalmic Solution for Treatment of Corneal Edema in Fuchs Dystrophy. Am J Ophthalmol. 2021 Jul;227:100-105. doi: 10.1016/j.ajo.2021.03.006. Epub 2021 Mar 15. PMID 33737034

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Netarsudil | Placebo
Started | 15 | 14
Completed | 13 | 13
Not Completed | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Netarsudil | Placebo | Total
Number analyzed (Participants) | 15 | 14 | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 68 (5) | 69 (7) | 68 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 9 | 18
  Male | 6 | 5 | 11
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White, non-Hispanic | 15 | 14 | 29
Region of Enrollment [Number; unit: participants]
  United States | 15 | 14 | 29

OUTCOME MEASURES:

1. Primary Outcome: Change in Central Corneal Thickness
Description: Central corneal thickness at 1 month after randomization minus central corneal thickness at baseline
Time Frame: 1 month
Measure: Mean (95% Confidence Interval); unit: microns
Arm/Group | Netarsudil | Placebo
Number analyzed (Participants) | 13 | 13
microns | -23 [-32 to -13] | -2 [-9 to 5]

2. Secondary Outcome: Change in Corrected Distance Visual Acuity (CDVA)
Description: Change in CDVA (lines read on the eye chart at 3 months minus lines read at baseline)
Time Frame: 3 months
Measure: Mean (95% Confidence Interval); unit: lines on the eye chart
Arm/Group | Netarsudil | Placebo
Number analyzed (Participants) | 13 | 13
lines on the eye chart | 1.9 [0.8 to 3] | 0.3 [-0.7 to 1.3]

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Netarsudil | Placebo
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/14
Other Adverse Events (participants affected / at risk) | 6/15 | 3/14
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Netarsudil (N=15) | Placebo (N=14)
conjunctival hyperemia (Eye disorders) | 6 (6) | 3 (3)
ocular irritation (Eye disorders) | 2 (2) | 1 (1)
glare (Eye disorders) | 1 (1) | 0 (0)
lacrimation (Eye disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-02-18): https://cdn.clinicaltrials.gov/large-docs/63/NCT04051463/Prot_SAP_000.pdf